CLINICAL TRIAL: NCT04478630
Title: The Effects of Inhaled Aromatherapy on Chemotherapy Induced Nausea and Vomiting (CINV) in Men and Women With Breast Cancer
Brief Title: The Effects of Inhaled Aromatherapy on Chemotherapy Induced Nausea (CINV) and Vomiting
Acronym: CINV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Doctors Kienle Center for Humanistic Medicine/Penn State College of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 19-104
Record Dates: First submitted 2020-07-07; First posted 2020-07-21 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: This study is a three group, randomized, double blind, placebo-controlled trial with two repeated measurements. The same measurements will be collected for each participant during two consecutive chemotherapy treatment cycles.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Subjects and all members of the research team will not know which group, either peppermint essential oil, ginger essential oil, or placebo (vanilla extract group), the potential subject would be randomly assigned to as the research team members involved in consenting will open a prefilled envelope to determine the group which will be labeled with the correlating diffuser (A, B, or C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peppermint Essential Oil (Active Comparator): Usual care plus a personal pocket diffuser prepared with 14 drops of peppermint essential oil. Each subject will be instructed to inhale from the pocket diffuser beginning on the day of their chemotherapy (Day 1) and continue using the inhaler for the next three consecutive days (Day 1-Day 4).The subjects will remove the cover of the pocket diffuser, place the pocket diffuser approximately an inch away from their nose and inhale three times with deep breathing (i.e., three sniffs). Subjects will take 3 sniffs of the aromatherapy inhaler three times daily (morning, afternoon, and evening).The subjects will complete a Pre-treatment Assessment form before cycle of chemotherapy (total of 2), as well as 24 and 72 hours after each cycle of chemotherapy. The exact same procedures will be repeated during the participant's next cycle of chemotherapy, which is likely two or three weeks after the first one.
  Interventions: Other: Peppermint Essential Oil, Ginger Essential Oil, or Pure Vanilla Extract
- Ginger Essential Oil (Active Comparator): Usual care plus a personal pocket diffuser prepared with 14 drops of ginger essential oil. Each subject will be instructed to inhale from the pocket diffuser beginning on the day of their chemotherapy (Day 1) and continue using the inhaler for the next three consecutive days (Day 1-Day 4). The subjects will remove the cover of the pocket diffuser, place the pocket diffuser approximately an inch away from their nose and inhale three times with deep breathing (i.e., three sniffs). Subjects will take 3 sniffs of the aromatherapy inhaler three times daily (morning, afternoon, and evening). The subjects will complete a Pre-treatment Assessment form before cycle of chemotherapy (total of 2), as well as 24 and 72 hours after each cycle of chemotherapy.The exact same procedures will be repeated during the participant's next cycle of chemotherapy, which is likely two or three weeks after the first one.
  Interventions: Other: Peppermint Essential Oil, Ginger Essential Oil, or Pure Vanilla Extract
- Pure Vanilla Extract (placebo-control) (Placebo Comparator): Usual care plus a personal pocket diffuser prepared with 14 drops of pure vanilla extract (placebo). Each subject will be instructed to inhale from the pocket diffuser beginning on the day of their chemotherapy (Day 1) and continue using the inhaler for the next three consecutive days (Day 1-Day 4). The subjects will remove the cover of the pocket diffuser, place the pocket diffuser approximately an inch away from their nose and inhale three times with deep breathing (i.e., three sniffs). Subjects will take 3 sniffs of the aromatherapy inhaler three times daily (morning, afternoon, and evening). The subjects will complete a Pre-treatment Assessment form before cycle of chemotherapy (total of 2), as well as 24 and 72 hours after each cycle of chemotherapy. The exact same procedures will be repeated during the participant's next cycle of chemotherapy, which is likely two or three weeks after the first one.
  Interventions: Other: Peppermint Essential Oil, Ginger Essential Oil, or Pure Vanilla Extract

INTERVENTIONS:
Other: Peppermint Essential Oil, Ginger Essential Oil, or Pure Vanilla Extract — Inhaled Aromatherapy via a pocket sized diffuser which contains one of the following:Peppermint Essential Oil, Ginger Essential Oil, or Pure Vanilla Extract (placebo-control).

SUMMARY:
This study is a three group, randomized, double blind, placebo-controlled trial with two repeated measurements. The same measurements will be collected for each participant during two consecutive chemotherapy treatment cycles.Subjects will be provided with written instructions as an educational handout as well as essential oil safety information. Subjects will be able to demonstrate an ability and accurate understanding of the proper use of the diffusers, using a demonstration diffuser, at the time of consent.

At the time the subject will provide written informed consent, they will be randomly assigned to one of the three groups with a pocket diffuser containing either ginger essential oil, peppermint essential oil, or vanilla extract )placebo- control). This is based on a pre-determined list of random assignments.

Each subject will be instructed to inhale from the pocket diffuser beginning on the day of their chemotherapy (Day 1) and continue using the inhaler for the next three consecutive days (Day 1-Day 4). The subjects will remove the cover of the pocket diffuser, place the pocket diffuser approximately an inch away from their nose and inhale three times with deep breathing (i.e., three sniffs). Subjects will take 3 sniffs of the aromatherapy inhaler three times daily (morning, afternoon, and evening).

In addition to the Pre-treatment Assessment, occurring before each of the 2 cycles of chemotherapy, the subjects will be contacted to complete assessments at approximately 24 and 72 hours post-chemotherapy. A member of the study team will call the participant again at their preferred time of day to ask the survey questions.

The same procedures will be repeated during the participant's second cycle of chemotherapy, which is likely two or three weeks after the first one.

DETAILED DESCRIPTION:
This study is a three group, randomized, double blind, placebo-controlled trial with two repeated measurements. The same measurements will be collected for each participant during two consecutive chemotherapy treatment cycles.

After subjects are identified to meet criteria and have reported some degree of nausea following chemotherapy, one of the Clinical Nurse Coordinators or Infusion Room Nurses on the research team will provide information regarding the study to the potential subject. If the potential subject is interested in participating in the study and physically demonstrates the ability to correctly use the pocket diffuser the consent will be gone over in detail with the potential subject and signed. Educational handouts outlining the instructions for use of the pocket diffuser as well as safety and contact information will be provided and explained to the subject at this time.

At the time the subject will provide written informed consent, they will be randomly assigned to one of the three groups (ginger essential oil, peppermint essential oil, or vanilla extract placebo- control) based on a pre-determined list of random assignments.

The diffusers will have been prepped with essential oils of either peppermint or ginger, which will each contain 14 drops of the designated essential oil. The nonessential oil diffusers (placebo) pure vanilla extract will also be prepared to each contain 14 drops each.

Prior to the start of the participant's chemotherapy infusion, all subjects will complete a pre-treatment survey to evaluate their baseline/anticipatory nausea. The pre-treatment survey will also include questions about the recent chemotherapy treatment experience related to appetite and the use of medication to prevent or lesson nausea.

Then, participants will be provided with their assigned pocket diffuser which has already been prepared with the correct substance (ginger essential oil, peppermint essential oil, or pure vanilla extract). Participants will be asked to remove the cover of the pocket diffuser, place the pocket diffuser about an inch under their nose, and inhale three times with deep breathing (i.e. three sniffs). After use, the inhaler should be capped to minimize dispersal of the scent. Subjects will take three sniffs of the aromatherapy inhaler three times daily (morning, afternoon, and evening) starting at the time of the chemotherapy appointment through the final survey at 72 hours post-discharge. Subjects will be instructed on proper disposal and receive a new pocket-sized diffuser at the next treatment visit.

All participants will be encouraged to follow all standard procedures related to their treatment including the use of any prescribed anti-emetics. Aromatherapy is considered a complementary therapy and is not intended to replace any current treatments.

During the day after chemotherapy administration (approximately 24 hours post-discharge), a member of the study team will call the participant at their preferred time of day to conduct the first post-intervention survey. This survey will be identical to the baseline survey conducted on Day 1, but it will also include questions about the aromatherapy diffuser usage. By calling 24 hours after chemotherapy, the nausea reported by the participant can be classified as "acute nausea." Additionally, it will be documented as to if the subject required any antiemetics in addition to what was planned and ordered per the standard chemotherapy regimen.

Approximately 72 hours post-discharge, a member of the study team will call the participant again at their preferred time of day. The survey questions will be exactly the same as the first phone call. At this time point, it will be possible to evaluate "delayed nausea" related to chemotherapy. Again, it will be documented as to if the subject required any antiemetics in addition to what was planned and ordered per the standard chemotherapy regimen.

Participants will be reminded during the call that they will receive a phone call from the study team prior to their next chemotherapy appointment to remind them to return their used pocket diffuser for disposal. Returning the used diffuser from the previous cycle will be helpful to ensure that the subject will not confuse the diffuser from the 1st and 2nd cycles. Although both diffusers will contain the same thing (ginger essential oil, peppermint essential oil, or pure vanilla extract), the used diffuser would be less potent as it has been opened multiple times.

The exact same procedures will be repeated during the participant's next cycle of chemotherapy, which is likely two or three weeks after the first one.

ELIGIBILITY:
Inclusion Criteria:

* Men and women included
* Ages between 21 years old and 89 years old
* Diagnosis of breast cancer - all histologies and stages
* Subjects must have reported some degree of nausea following chemotherapy
* Subjects must have at least two remaining cycles of chemotherapy to complete
* Subjects must be fluent in English or Spanish
* Subjects must be willing to complete questionnaire through follow-up phone calls
* Subjects must be able to use the pocket diffuser

Exclusion Criteria:

* Inability to sign the consent
* Pregnancy
* Cognitive impairment
* Current use of aromatherapy for symptom management or prevention
* Allergies to peppermint, ginger, or vanilla
* Concurrent radiation therapy

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-02-18 (Actual)

PRIMARY OUTCOMES:
Acute Nausea Score | 24 hours post-chemotherapy
  N&V experienced during the first 24 hours after chemotherapy administration as measured by the Memorial Symptom Assessment Scale's nausea and vomiting dimension with values for symptoms, if experienced, on a 4-point scale; its frequency, if appropriate, on a 4-point scale; and its associated distress on a 5-point categorical scale. The higher the score determines a worse outcome in all areas.
Delayed Nausea Score | 72 hours post-chemotherapy
  N&V that occurs more than 24 hours after chemotherapy administration , as measured by the Memorial Symptom Assessment Scale's nausea and vomiting dimension, with values for symptoms, if experienced, on a 4-point scale; its frequency, if appropriate, on a 4-point scale; and its associated distress on a 5-point categorical scale. The higher the score determines a worse outcome in all areas.

SECONDARY OUTCOMES:
Appetite For the 24 Hours Post-chemotherapy | 24 hours post-chemotherapy
  Approximately 24 hours after chemotherapy administration, a member of the study team will call the participant at their preferred time of day to conduct a post-chemotherapy survey and include documentation of the questions regarding appetite: ability to eat as they normally would, less than they normally would eat, no appetite, or inability to eat most foods.
Appetite During the 72 Hours Post-chemotherapy | 72 hours post-chemotherapy
  Approximately 72 hours after chemotherapy administration, a member of the study team will call the participant at their preferred time of day to conduct a post-chemotherapy survey and include documentation of the questions regarding appetite: ability to eat as they normally would, less than they normally would eat, no appetite, or inability to eat most foods.
Use of additional anti-emetic medications (in addition to the standard regimen's listed anti-emetics) | 24 hours post-chemotherapy
  Approximately 24 hours after chemotherapy administration, a member of the study team will call the participant at their preferred time of day to conduct a post-chemotherapy survey and include documentation of the name and frequency of any anti-emetics used in addition to the standard regimen's anti-emetics.
Use of additional anti-emetic medications (in addition to the standard regimen's listed anti-emetics) | 72 hours post-chemotherapy
  Approximately 72 hours after chemotherapy administration, a member of the study team will call the participant at their preferred time of day to conduct a post-chemotherapy survey and include documentation of the name and frequency of any anti-emetics used in addition to the standard regimen's anti-emetics.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The Clinical Study Report will be available to other researchers after the study and data are finalized.
Supporting Information: CSR
Time Frame: The data will become available after the study results are finalized. This is estimated to occur December 2020.